CLINICAL TRIAL: NCT07388433
Title: Exploring Behavioral Interventions to Improve Adherence to Multiple Micronutrient Supplements Among Pregnant Women in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller International (Other)
Collaborators: University of British Columbia (Other); Minstry of Health of Cambodia, National Maternal and Child Health Center (Unknown); Ministry of Health of Cambodia, National Nutrition Program (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: NECHR No. 346
Record Dates: First submitted 2026-01-09; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Adherence to Care
Keywords: multiple micronutrient supplements; pregnancy; adherence; implementation science; Cambodia; behavior change; COM-B model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Support Session; Tracking Calendar, and MMS eduational video package (Experimental): Single cohort of pregnant women receiving multiple micronutrient supplements throughout pregnancy plus sequential exposure to three behavioral interventions (family support session, tracking calendar, and educational SMS-style videos) to support daily MMS adherence and healthy pregnancy practices.
  Interventions: Behavioral: Family support session; Behavioral: Tracking Calendar; Behavioral: MMS educational video package

INTERVENTIONS:
Behavioral: Family support session — One 1 hour group session at the health center in Khmer for each participant and two self selected family members, facilitated by trained midwives and research staff, covering antenatal care, importance of daily MMS, and specific actions family members can take (reminders, workload support, healthy behaviors); includes interactive discussion and a summary handout for each family member.
Behavioral: Tracking Calendar — Culturally tailored wall calendar designed by a social marketing group, pretested with pregnant women, with daily visual tick boxes to mark MMS intake, reminders for ANC visits, and illustrated messages on recommended and discouraged pregnancy behaviors; provided with in person orientation on use and kept at home for at least 3 weeks.
Behavioral: MMS educational video package — Three short Khmer language videos (one per week over 3 weeks) sent via Telegram, featuring midwives providing counseling on daily MMS, managing side effects, healthy pregnancy practices, and the role of family support; scripts developed by the research team and maternal health experts and pretested with pregnant women.

SUMMARY:
The goal of this mixed method study is to learn how three different behavioral interventions can help pregnant women in Cambodia take a daily multiple micronutrient supplement (MMS) as recommended during pregnancy and to understand how acceptable and useful these interventions are for them. The main questions it aims to answer are:

* How do family support sessions, a tracking calendar, and short educational videos help pregnant women remember to take MMS every day and follow healthy pregnancy practices?
* Which of these three interventions do pregnant women find most helpful and acceptable for supporting daily MMS use?

Researchers will compare the three interventions (family support, tracking calendar, and educational videos) to see which approach best supports high MMS adherence and is most preferred by pregnant women.

Participants will:

* Take MMS tablets every day during pregnancy, starting from early pregnancy.
* Invite two family members to attend a one-hour group session at the health center about MMS and healthy pregnancy, including how families can support daily supplement use.
* Use a culturally tailored tracking calendar at home for three weeks to mark each day they take MMS and see reminders about clinic visits and healthy pregnancy behaviors.
* Receive one short motivational video per week for three weeks via Telegram, featuring midwives who explain MMS, answer common concerns, and encourage daily supplement use.
* Join focus group discussions after each intervention to share their experiences, preferences, and suggestions, and have remaining tablets counted to measure how many doses they took.

DETAILED DESCRIPTION:
This mixed-methods study will explore how three behavioral interventions can support pregnant women in Cambodia to take a daily multiple micronutrient supplement (MMS) as recommended throughout pregnancy and how acceptable and useful these interventions are in their daily lives. The study is being conducted in four provinces in Cambodia (Kampong Chhnang, Ratanakiri, Takeo, and Kampot) and enrolls healthy pregnant women in early pregnancy who attend antenatal care (ANC) at selected health centers. Its findings will help inform Cambodia's planned transition from iron-folic acid to MMS by identifying feasible, family- and community-appropriate strategies to promote high adherence.

The study focuses on three behavioral interventions: (1) a family support session, (2) a tracking calendar, and (3) short educational videos delivered via mobile phone. All enrolled participants are asked to take MMS daily and are sequentially exposed to each of the three interventions, with time between them to try out and reflect on each one. After using each intervention for approximately three weeks, participants join a focus group discussion to describe their experiences, including what helped or hindered their daily MMS intake and what they liked or disliked about the intervention. At each discussion, study staff also count remaining MMS tablets to calculate adherence over that period.

The family support intervention is designed to strengthen the role of close relatives-especially husbands and other key family members-in supporting women's daily MMS intake and broader healthy pregnancy practices. Each pregnant woman is invited to bring two family members of her choice to a one-hour, group-based session at the health center, led by trained midwives and research staff. The session covers essential ANC topics, the benefits and importance of daily MMS, and specific, practical ways family members can help, such as giving reminders, reducing the woman's household workload, or helping her keep MMS in a visible place. Family members can ask questions, discuss challenges, and receive a take-home handout summarizing key messages and suggested supportive actions. Women then return home and experience family support in their everyday context for about three weeks before attending a focus group discussion to describe what kind of support they actually received and how it affected their MMS-taking routine.

The tracking calendar intervention provides a visual tool that women can use at home to monitor and encourage their daily MMS intake and healthy pregnancy behaviors. After completing the family support phase, each participant receives a culturally tailored calendar designed with simple Khmer text and clear illustrations that are suitable for users with varying literacy levels. The calendar includes a daily space to mark when MMS has been taken, reminders for scheduled ANC visits, and icons that promote positive pregnancy practices such as eating a balanced diet and resting, as well as icons indicating behaviors to avoid, such as alcohol use and heavy lifting. Research staff give a short orientation on how to use the calendar, showing women how to mark each day and interpret the symbols. Women then use the calendar at home for about three weeks. A follow-up focus group discussion is conducted to learn how they used the calendar, whether it helped them remember to take MMS, what they found easy or difficult, and what improvements they suggest.

The video intervention uses digital communication to reach women in their homes and reinforce key MMS and pregnancy messages. Over a three-week period, participants receive one short motivational video per week via Telegram, a commonly used messaging application in Cambodia. The videos are in Khmer and feature midwives providing counseling and encouragement on daily MMS adherence, addressing common reasons for missed doses (such as forgetfulness or side effects), and emphasizing the importance of family support. The scripts are developed by the research team with input from maternal health experts, and the videos are pretested with pregnant women not enrolled in the main study to ensure that the messages are clear, relevant, and engaging. At the end of the three-week video period, participants take part in another focus group discussion to share how they watched and understood the videos, what they found most useful or challenging, and whether the videos influenced their MMS-taking habits.

Across all intervention periods, the study team collects both qualitative and quantitative data. Qualitative data come from focus group discussions conducted in Khmer at health centers, using semi-structured guides that explore participants' perceptions of relevance, acceptability, ease of use, and perceived impact of each intervention on MMS adherence and broader pregnancy behaviors. Discussions are audio-recorded and transcribed verbatim in Khmer, then translated into English for analysis by a trained research team using a structured content analysis approach informed by the COM-B (Capability, Opportunity, Motivation-Behavior) model. This framework helps identify how knowledge, practical skills, social support, and motivation influence women's ability to take MMS every day. Quantitative data include sociodemographic characteristics collected at enrollment, pill counts after each intervention period to objectively measure adherence, and an MMS acceptability survey administered using a Likert-scale questionnaire that covers taste, packaging, burden, perceived effectiveness, opportunity cost, and self-efficacy.

Eligible participants are pregnant individuals aged 18 to 45 years, in their first 14 weeks of a low-risk, singleton pregnancy, attending their first ANC visit at one of the participating health centers, living in one of the four study provinces with no plan to relocate within the next four months, willing to take MMS as their prenatal supplement, and able to participate in three focus group discussions. Women with high-risk pregnancies or plans to move away during the study period are excluded. The anticipated sample size is 36 enrolled pregnant women (approximately 9 per province), with the expectation that some may be unable to attend all focus group sessions due to relocation, work, or pregnancy-related events. All participants receive MMS following the UNIMMAP formulation and are asked to take one tablet per day throughout the study.

The main outcomes of interest are: (1) women's perceptions of the acceptability, relevance, and usefulness of each behavioral intervention for supporting MMS adherence and healthy pregnancy practices; (2) participants' preferences and rankings of the three interventions based on their experiences; and (3) adherence to MMS as measured by pill counts during each intervention period. Secondary outcomes include women's suggestions for improving the content and delivery of future MMS adherence interventions; descriptions of how family members, social environments, and daily routines influence MMS use; and quantitative measures of MMS acceptability across several domains. These findings will provide practical guidance for Cambodian health authorities and partners on how to design and scale effective behavioral strategies that can be integrated into ANC services and community-based programming as MMS is rolled out nationally.

ELIGIBILITY:
Inclusion Criteria:

* 14 weeks' gestation at first ANC visit (low risk, singleton pregnancy)
* Attending first ANC visit at one of the participating health centers in Kampong Chhnang, Ratanakiri, Takeo, or Kampot
* Residing in one of the four study provinces with no plans to relocate in the next 4 months
* Willing to take MMS as prenatal supplement for the study period
* Willing to participate in three focus group discussions (plus final ranking discussion)

Exclusion Criteria:

* Pregnancy classified as high risk by the healthcare provider (any medical condition that makes pregnancy high risk)
* Plan to relocate outside the four study provinces within 4 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-identified women who are currently pregnant and meet all other eligibility criteria are eligible to participate.
Enrollment: 36 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
COM-B-based qualitative themes on determinants of MMS adherence | 3-4 weeks after starting each new intervention
  Thematic analysis (content analysis) of FGD transcripts mapped onto COM B domains (capability, opportunity, motivation) to identify perceived barriers and facilitators related to each intervention and MMS adherence.
Participant ranking of three behavioral interventions for supporting MMS adherence | At endline or approximately 90 days after enrollment, following completion of all three interventions.
  Participants rank family support, tracking calendar, and educational videos from 1 (most effective) to 3 (least effective) in supporting daily MMS adherence and healthy pregnancy practices; rankings summarized descriptively overall and by province.

OTHER OUTCOMES:
MMS adherence (%) over the intervention period | 3-4 weeks from start of each intervention
  Proportion of prescribed MMS tablets consumed, calculated as the number of tablets taken divided by the number of tablets eligible to be consumed between the first ANC visit and the pill count; measured via direct tablet counts at the end of each 3-week intervention period.
Acceptability of MMS and behavioral interventions | At endline or approximately 90 days after enrollment, following completion of all three interventions.
  Participant-reported acceptability across domains: physical properties, packaging, burden, perceived effectiveness, opportunity cost, and self-efficacy using an interviewer-administered Likert scale questionnaire; acceptability summarized as proportion agreeing or strongly agreeing with positive statements.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh Hoang, Master of Public Health, Principal Investigator — Helen Keller Intl; Kim Rattana, Medical Doctor, Study Chair — Minstry of Health of Cambodia, National Maternal and Child Health Center
Locations (1):
- Prey Khmer Health Center in Kampong Chhnang; Prambei Mom Health Center in Takeo Province; Chakrey Ting Health Center in Kampot Province; Kon Mon Health Center in Ratanakiri Province, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Undecided
A decision on sharing (PD has not yet been made because the study's current ethics approval from the National Ethics Committee for Health Research (NECHR) in Cambodia does not explicitly cover IPD sharing outside the primary research team. Before any IPD could be shared, additional approval or guidance from NECHR would be required to ensure full protection of participant privacy and compliance with national ethical and regulatory requirements.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT07388433/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT07388433/ICF_001.pdf